CLINICAL TRIAL: NCT02099188
Title: Multidisciplinary Approach for Poor Prognosis Sinonasal Tumors: Phase II Study of Chemotherapy, Photon and Heavy Ion Radiotherapy Integration for More Effective and Less Toxic Treatment in Inoperable Patients
Brief Title: Multidisciplinary Approach for Poor Prognosis Sinonasal Tumors in Inoperable Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Regione Lombardia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINTART2; 2013-000580-93 (EudraCT Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-28 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2022-04

CONDITIONS: Unresectable Sinonasal Tumors
MeSH Terms: interventions — Cisplatin; Docetaxel; Fluorouracil; Etoposide; Doxorubicin; Ifosfamide; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multimodality treatment (Experimental): Squamocellular Carcinoma, Sinonasal Undifferentiated Carcinoma:
  * Docetaxel at 75 mg/m2 as IV infusion on Day 1 q3w
  * Cisplatin at 80 mg/m2 as IV infusion on Day 1 q3w
  * 5-fluorouracil at 800 mg/m2/day as IV infusion from Day 1 to Day 4 q3w
  Small cell carcinoma neuroendocrine type, Pure neuroendocrine carcinoma and grade III-IV Esthesioneuroblastoma.
  * Cisplatin at 33 mg/m2/day as IV infusion from Day 1 to Day 3 q3w.
  * Etoposide at 150 mg/m2/day as IV infusion from Day 1 to Day 3 q3w . Second cycle and every other cycle
  * Adriamycin at 20 mg/m2/day as IV infusion from Day 1 to Day 3 q3w.
  * Ifosfamide at 3000 mg/m2/day as IV infusion from Day 1 to Day 3 q3w.
  Intestinal Type Adenocarcinoma with functional p53.
  * Leucovorin* at 250 mg/m2/day as IV infusion from Day 1 to Day 5 q3w.
  * Cisplatin at 100 mg/m2 as IV infusion on Day 2 q3w
  * 5-fluorouracil at 800 mg/m2/day as IV infusion from Day 2 to Day 5 q3w
  Followed by radiotherapy
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: 5-fluorouracil; Drug: Etoposide; Drug: Adriamycin; Drug: Ifosfamide; Drug: Leucovorin; Radiation: Radiotherapy - Patients needing Elective Nodal Volume (ENI); Radiation: Radiotherapy - Patients not needing ENI; Radiation: Radiotherapy - Patients needing curative neck irradiation

INTERVENTIONS:
Drug: Cisplatin — 80 mg/m2 or 33 mg/m2/day or 100 mg/m2 - Concentrate for solution for infusion
  Other Names: CDDP
Drug: Docetaxel — 75 mg/m2 - Concentrate for solution for infusion
  Other Names: Taxotere
Drug: 5-fluorouracil — 800 mg/m2/day - Concentrate for solution for infusion
  Other Names: Adrucil
Drug: Etoposide — 150 mg/m2/day - Concentrate for solution for infusion
  Other Names: Vepesid
Drug: Adriamycin — 20 mg/m2/day - Powder for solution for infusion
  Other Names: Doxorubicin
Drug: Ifosfamide — 3000 mg/m2/day - Powder for solution for infusion
  Other Names: Ifex
Drug: Leucovorin — 250 mg/m2/day - Powder for solution for infusion
  Other Names: Folinic acid
Radiation: Radiotherapy - Patients needing Elective Nodal Volume (ENI) — LR-PTV: 50.4-54 Gy with 1.8-2 Gy per fraction will be prescribed. This volume will always be treated with photons IMRT.
  1. Particle boost with ENI:
     HR-PTV: carbon ions 18 - 21 Gy (relative biological effectiveness, RBE) in fractions of 3 Gy (RBE) without concomitant chemotherapy IR-PTV: this volume is optional, if used it will receive the first 3 fractions i.e. 9 Gy (RBE) of the boost.
  2. Photons boost with ENI. HR-PTV: at least 70 Gy with 2-2.12 Gy per fraction and 66 Gy at 2Gy per fraction in radical setting will be prescribed. IR-PTV: 59.4-60 Gy with 1.8 Gy-2 Gy per fraction will be prescribed.
Radiation: Radiotherapy - Patients not needing ENI — 1. Treatment with particles. IR-PTV: this volume can be larger or equal to HR-PTV according to individual situations. 50.4-54 Gy with 1.8-2 Gy per fraction will be prescribed to IR-PTV with protontherapy with concomitant chemotherapy. HR-PTV: carbon ions 18 - 21 Gy (RBE) in fractions of 3 Gy (RBE) without concomitant chemotherapy. The first 3 fractions may be given to the bigger IR-PTV.
  2. Treatment with photons. HR-PTV: at least 70 Gy with 2-2.12 Gy per fraction and 66 Gy at 2Gy per fraction in radical setting will be prescribed. IR-PTV: 59.4-60 Gy with 1.8 Gy-2 Gy per fraction will be prescribed.
Radiation: Radiotherapy - Patients needing curative neck irradiation — LR-PTV: 50.4-54 Gy with 1.8-2 Gy per fraction will be prescribed. This volume will always be treated with photons IMRT.
  1. Particle boost. HR-PTV: carbon ions 18 - 21 Gy (RBE) in fractions of 3 Gy (RBE) without concomitant chemotherapy IR-PTV: this volume is optional, if used it will receive the first 3 fractions i.e. 9 Gy (RBE) of the boost.
  2. Photons boost. HR-PTV: at least 70 Gy with 2-2.12 Gy per fraction and 66 Gy at 2Gy per fraction in radical and postoperative setting will be prescribed. IR-PTV: 59.4-60 Gy with 1.8 Gy-2 Gy per fraction will be prescribed.

SUMMARY:
Sinonasal tumors are rare diseases, as they account for the 0.2 % - 0.8 % of all tumors. For patients with inoperable tumors, the prognosis is poor and the current therapy is a combined-modality treatment that is both more effective and associated with less morbidity.

This study proposes innovative integration of multiple modality of treatment modulated by histology, molecular profile and response to induction CT.

DETAILED DESCRIPTION:
So far, surgery followed by radiotherapy (RT) has been the usual approach for advanced disease. Technical improvements in surgical approaches have been reported, providing less invasive surgery with lower morbidity. However, there are cases of unresectable tumors where the needs of novel strategies is higher.

New therapeutic strategies are needed to obtain more efficient treatment with less morbidity. Some studies explored the role and feasibility of induction chemotherapy (CT) and the prognostic value of response to CT. Histology and molecular pattern can guide the type of administered CT. The first drives the choice of drug to be associated with Cisplatin, while mutational status of p53 (wild type, WT vs mutated, MUT) is a predictive value for response to CT with Cisplatin plus 5-Fluorouracil and Leucovorin in ITAC.

Moreover, proton/carbon ion beam therapy, compared to conventional photon therapy, provides a more accurate and intense dose to tumor area, with potentially higher control of disease.

Treatment outcomes for unresectable paranasal sinus carcinoma are poor, and combined-modality treatment is needed to find out novel therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated IEC-approved Informed Consent.
2. Diagnosis of sinonasal tumor with the following histotypes:

   * Squamous Cell Carcinoma (SCC);
   * Sinonasal Undifferentiated Carcinoma (SNUC);
   * Small Cell Carcinoma Neuroendocrine Type (SmCCNET);
   * Pure Sinonasal Neuroendocrine Carcinoma (SNEC);
   * Intestinal Type Adenocarcinoma (ITAC) with a functional p53 gene;
   * Esthesioneuroblastoma with differentiation grade III-IV by Hyams.
3. AJCC stage T4b.
4. Unresectable disease.
5. ECOG performance status 0-2.
6. Adequate bone marrow, renal and hepatic functionality, defined as haemoglobin >10 g/dL, neutrophils >1500/mmc, platelets > 100.000/mmc, creatinine value ≤ 1.5 x ULN or calculated creatinine clearance (by Cockcroft and Gault's formula) > 60 mL/min, transaminases values < 1.5 times over the upper limit of normal (ULN).
7. Polychemotherapy treatment clinical feasibility as per Investigator's Judgment.
8. Male or female patients ≥ 18 years of age.
9. Negative pregnancy test (if female in reproductive years).
10. Agreement upon the use of effective contraceptive methods (hormonal or barrier method of birth control, or abstinence) prior to study entry and for the duration of study participation, if men and women of child producing potential.

Exclusion Criteria:

1. Previous radiotherapy or chemotherapy for head and neck district tumors (surgical treatment relapses are admitted).
2. Metastatic disease.
3. Cardiac, pulmonary, infective, neurological disease or any other medical condition that could interfere with treatment.
4. Unable and unwilling to comply with scheduled visits, therapy plans, and laboratory tests required in this protocol.
5. Previous diagnosis of other malignant neoplasm in the last 3 years (in situ cervical cancer or completely excised basocellular/squamocellular skin cancer are always admitted).
6. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11; Primary Completion 2020-06 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | PFS will be assessed at 5 years.
  Progression Free Survival (PFS) at 5 years, defined as the time from enrollment to progression of disease or death for any cause; last date of follow up will be registered for patients alive not in progression.

SECONDARY OUTCOMES:
Overall survival (OS) | Overall survival will be assessed at the following time frames: 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months.
  Overall survival defined as the time from enrollment (ITT population) or treatment start (PP population) to the date of death from any causes; last date of follow up will be registered for patients alive.
Ocular function preservation by visual field tests. | At the enrollment. During follow-up after: 3 months, 12 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months.
  Ocular function preservation by visual field tests.
Hearing preservation performed by audiogram test. | At the enrollment. During follow-up after: 3 months, 12 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months.
  Hearing preservation performed by audiogram test.
Overall safety profile of the whole treatment. | From the day of the Informed Consent Form signature through to 90 days after the last dose of the last therapy administered (i.e., radiotherapy and/or chemotherapy).
  Overall safety profile of the whole treatment characterized by type, severity graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4.03), timing and relationship to study therapy of adverse events and laboratory abnormalities collected.
Objective Response Rate | After the end of 1st, 3rd and 5th cycle of induction therapy and before the radiotherapy. During f-up at the following time frames: 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months, 60 months.
  Objective Response Rate (CR and PR by RECIST criteria version 1.1)
Adverse events and laboratories abnormalities. | During the treatments. F-up at the following time frames: 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months.
  Adverse events (characterized by type, severity, timing) and laboratories abnormalities (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4.03), induced by radiotherapy (both photon RT and heavy ion RT).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Study Director — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI; Piero Nicolai, MD, Principal Investigator — Presidi Ospedalieri Spedali Civili di Brescia; Paolo Castelnuovo, MD, Principal Investigator — A.O. Ospedale di Circolo e Fondazione Macchi; Marco Benazzo, MD, Principal Investigator — IRCCS Policlinico San Matteo; Letizia Deantonio, MD, Principal Investigator — Azienda Ospedaliera "Maggiore della Carità"
Locations (5):
- Italy (5):
  - Presidio Ospedaliero Spedali Civili di Brescia, Brescia, BS
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan, MI
  - IRCCS Policlinico San Matteo, Pavia, PV
  - A.O. Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Azienda Ospedaliera "Maggiore della Carità", Novara